CLINICAL TRIAL: NCT00930137
Title: Ruminant Trans Fats and the Risk of Cardiovascular Disease in Women
Acronym: TRANSW
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Laval University (Other)
Collaborators: Institute of Nutraceuticals and Functional Foods (Other); Dairy Farmers of Canada (Other); Dairy Australia (Industry)
Responsible Party: Principal Investigator, Benoit Lamarche, Professor, Laval University
Allocation: Randomized | Model: Crossover | Masking: Quadruple | Purpose: Prevention
Other Study IDs: INAF-2009-084
Record Dates: First submitted 2009-06-29; First posted 2009-06-30 (Estimated); Last update posted 2013-03-05 (Estimated); Status verified 2013-03

CONDITIONS: Cardiovascular Disease
Keywords: Cardiovascular disease; Trans fatty acids; Ruminant; Blood lipids; Lipoproteins; Women
MeSH Terms: conditions — Cardiovascular Diseases

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (2):
- High dairy trans fat (Experimental): a diet rich in ruminant trans fatty acids (4.1 g/2500 kcal)
  Interventions: Other: isocaloric for week diet
- Low dairy trans fat diet (Active Comparator): a control diet (minimal dietary ruminant trans fatty acids, 0.7 g/2500 kcal)
  Interventions: Other: isocaloric for week diet

INTERVENTIONS:
Other: isocaloric for week diet — Consumption of the 2 experimental diets
  1. a diet rich in ruminant trans fatty acids (4.1 g/2500 kcal);
  2. a control diet (minimal dietary ruminant trans fatty acids, 0.7 g/2500 kcal).

SUMMARY:
While the deleterious effects of trans fat from industrial sources (iTFA) on cardiovascular health are well established, the impact of TFA from ruminants (rTFA) on cardiovascular risk factors has not been as well characterized. We have previously shown in men that a very high dietary intakes of rTFA (>3.5% of energy) leads to unfavourable changes in lipid cardiovascular risk factors that are similar to those seen with iTFA. However, our data also indicated that achievable intakes of rTFA that remain well above the current human consumption (1.5% of energy intake) had neutral effects on plasma lipids and other cardiovascular disease (CVD) risk factors in men. Other studies have also suggested that the LDL and HDL response to very high dietary intakes of rTFA (>5% of energy) in women may be different than in men.

The general objective of the study is to investigate for the first time in a double-blind randomized controlled study the impact of high but yet achievable intake of ruminant trans fatty acids on plasma LDL-Cholesterol and other risk factors for CVD in healthy women.

DETAILED DESCRIPTION:
Ruminant trans fatty acids (rTFA) will come from an experimental butter formulated from dairy fat obtained after having modified the regimen of lactating cows. All diets will be identical in terms of menus, calories and macronutrient composition with the exception of TFA levels. All foods will be provided to study participants. Based on a 2500 kcal/day regimen, an intake of 4.1g of rTFA will represent 37 kcal/day (1.5% of energy intake) while the intake of 0.7 g of rTFA in the control diet will represent 6 calories (0.3% of energy). The 2 experimental diets will be formulated so that the percentage of daily calories from fat (33%), carbohydrates (52%) and proteins (15%) will meet the dietary recommendations of the American Heart Association and the NCEP for primary prevention of CVD.

ELIGIBILITY:
Inclusion Criteria:

* Healthy women using or not contraceptive agents or hormone supplementation
* For pre-menopausal women: regular menstrual cycle for the last 3 months (25- 35 days)
* LDL-Cholesterol concentration between 2.5 and 4.0 mmol/L
* Stable body weight (+/- 2 kg) for 6 months before the beginning of the study
* Smoking or not

Exclusion Criteria:

* Previous history of cardiovascular disease, type 2 diabetes and monogenic dyslipidemia
* Subjects taking medications for hyperlipidemia or hypertension
* Endocrine disorders
* Body mass index > 35 kg/m2
* Food allergies
* Women with extreme nutritional habits such as vegetarism or alcohol consumption > 2 drinks/day
* Elite athletes

Ages: 18 Years to 70 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 64 (Actual)
Dates: Start 2009-09; Primary Completion 2010-12 (Actual); Study Completion 2011-09 (Actual)

PRIMARY OUTCOMES:
Plasma LDL-Cholesterol concentrations | At the beginning of the study and the end of the 2 for-week diets

SECONDARY OUTCOMES:
Blood lipids and apolipoproteins (Total cholesterol, HDL-Cholesterol, Triglycerides, Apo A1, Apo B) | At the beginning of the study and the end of the 2 for-week diets
CRP | At the beginning of the study and the end of the 2 for-week diets
Blood pressure | At the beginning of the study and the end of the 2 for-week diets
Anthropometric measures (waist and hip circumferences) | At the beginning of the study and the end of the 2 for-week diets

CONTACTS AND LOCATIONS:
Overall Officials: Benoît Lamarche, PhD, Principal Investigator — Institute of Nutraceutical and Functional Foods (INAF), Laval University; Patrick Couture, MD, FRCP (C, PhD), Study Director — Faculty of Medicine, Laval University
Locations (1):
- Institute of Nutraceutical and Functional Foods (INAF), Laval University, Québec, Quebec, Canada

REFERENCES:
- [Background] Motard-Belanger A, Charest A, Grenier G, Paquin P, Chouinard Y, Lemieux S, Couture P, Lamarche B. Study of the effect of trans fatty acids from ruminants on blood lipids and other risk factors for cardiovascular disease. Am J Clin Nutr. 2008 Mar;87(3):593-9. doi: 10.1093/ajcn/87.3.593. PMID 18326596
- [Background] Desroches S, Chouinard PY, Galibois I, Corneau L, Delisle J, Lamarche B, Couture P, Bergeron N. Lack of effect of dietary conjugated linoleic acids naturally incorporated into butter on the lipid profile and body composition of overweight and obese men. Am J Clin Nutr. 2005 Aug;82(2):309-19. doi: 10.1093/ajcn.82.2.309. PMID 16087973
- [Background] Mauger JF, Lichtenstein AH, Ausman LM, Jalbert SM, Jauhiainen M, Ehnholm C, Lamarche B. Effect of different forms of dietary hydrogenated fats on LDL particle size. Am J Clin Nutr. 2003 Sep;78(3):370-5. doi: 10.1093/ajcn/78.3.370. PMID 12936917
- [Background] Lichtenstein AH, Ausman LM, Jalbert SM, Schaefer EJ. Effects of different forms of dietary hydrogenated fats on serum lipoprotein cholesterol levels. N Engl J Med. 1999 Jun 24;340(25):1933-40. doi: 10.1056/NEJM199906243402501. PMID 10379016
- [Background] Chardigny JM, Destaillats F, Malpuech-Brugere C, Moulin J, Bauman DE, Lock AL, Barbano DM, Mensink RP, Bezelgues JB, Chaumont P, Combe N, Cristiani I, Joffre F, German JB, Dionisi F, Boirie Y, Sebedio JL. Do trans fatty acids from industrially produced sources and from natural sources have the same effect on cardiovascular disease risk factors in healthy subjects? Results of the trans Fatty Acids Collaboration (TRANSFACT) study. Am J Clin Nutr. 2008 Mar;87(3):558-66. doi: 10.1093/ajcn/87.3.558. PMID 18326592
- [Background] Tholstrup T, Raff M, Basu S, Nonboe P, Sejrsen K, Straarup EM. Effects of butter high in ruminant trans and monounsaturated fatty acids on lipoproteins, incorporation of fatty acids into lipid classes, plasma C-reactive protein, oxidative stress, hemostatic variables, and insulin in healthy young men. Am J Clin Nutr. 2006 Feb;83(2):237-43. doi: 10.1093/ajcn/83.2.237. PMID 16469980
- [Background] Oomen CM, Ocke MC, Feskens EJ, van Erp-Baart MA, Kok FJ, Kromhout D. Association between trans fatty acid intake and 10-year risk of coronary heart disease in the Zutphen Elderly Study: a prospective population-based study. Lancet. 2001 Mar 10;357(9258):746-51. doi: 10.1016/s0140-6736(00)04166-0. PMID 11253967
- [Background] Mozaffarian D, Katan MB, Ascherio A, Stampfer MJ, Willett WC. Trans fatty acids and cardiovascular disease. N Engl J Med. 2006 Apr 13;354(15):1601-13. doi: 10.1056/NEJMra054035. No abstract available. PMID 16611951
- [Background] Willett WC, Stampfer MJ, Manson JE, Colditz GA, Speizer FE, Rosner BA, Sampson LA, Hennekens CH. Intake of trans fatty acids and risk of coronary heart disease among women. Lancet. 1993 Mar 6;341(8845):581-5. doi: 10.1016/0140-6736(93)90350-p. PMID 8094827
- [Background] Willett W, Mozaffarian D. Ruminant or industrial sources of trans fatty acids: public health issue or food label skirmish? Am J Clin Nutr. 2008 Mar;87(3):515-6. doi: 10.1093/ajcn/87.3.515. No abstract available. PMID 18326587
- [Derived] Lacroix E, Charest A, Cyr A, Baril-Gravel L, Lebeuf Y, Paquin P, Chouinard PY, Couture P, Lamarche B. Randomized controlled study of the effect of a butter naturally enriched in trans fatty acids on blood lipids in healthy women. Am J Clin Nutr. 2012 Feb;95(2):318-25. doi: 10.3945/ajcn.111.023408. Epub 2011 Dec 28. PMID 22205319